CLINICAL TRIAL: NCT00953615
Title: Open Label, Phase II Investigation of Thalidomide for the Treatment of Primary Sclerosing Cholangitis
Brief Title: Thalidomide for the Treatment of Primary Sclerosing Cholangitis (PSC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Dr. K. Lindor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 342-06
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC; Thalidomide
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide (Experimental): Participants will be treated with Thalidomide, starting at a dose of 100 mg per day, increasing the dose by 100 mg every 14 days to a maximum of 400 mg per day.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Titrate to 400 mg daily for 6 months
  Other Names: Thalomid

SUMMARY:
The purpose of this study is to determine the safety and benefit of Thalidomide with primary sclerosing cholangitis (PSC). This is a six month study.

DETAILED DESCRIPTION:
At entry, patients will have a complete history and physical, blood tests, ultrasound, and will complete questionnaires. Eligible patients will take Thalidomide 400 mg once a day in the evening. Patients will start a dose of 100 mg per day for two weeks, increasing by 100 mg per day every two weeks to a maximum dose of 400 mg per day for 6 months. Patients will return at 6 months for an evaluation, blood tests and completion of questionnaires. Blood tests will be performed by mailed-in kits at 3 months. Patients will receive weekly phone calls for the first 2 months and bi-monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of primary sclerosing cholangitis as defined by: serum alkaline phosphatase level greater than or equal to 1.5 times the upper limit of normal, negative serum antimitochondrial antibody test, cholangiography diagnostic of PSC without other etiology for biliary obstruction, and liver histology consistent with or diagnostic of PSC
* Patients must give written informed consent.
* Patients must be willing and able to comply with the most recent version of the FDA-mandated System for Thalidomide Education and Prescribing Safety (S.T.E.P.S.®) program.

Exclusion Criteria:

* Pregnant and/or lactating female
* Inability or unwillingness to practice contraceptive measures for the prevention of pregnancy
* History of hypersensitivity reaction to thalidomide
* Inability to provide consent
* Findings suggestive of liver disease of other etiology such as primary biliary cirrhosis, chronic alcoholic liver disease, chronic hepatitis B and C infection, hemochromatosis, Wilson's disease, alpha-1-antitrypsin deficiency, autoimmune hepatitis, and cryptogenic liver disease
* Anticipated need for liver transplantation in one year from decompensated chronic liver disease or recurrent variceal bleeding, spontaneous hepatic encephalopathy, or refractory ascites
* Treatment with tacrolimus, cyclosporine, sirolimus, ursodeoxycholic acid, corticosteroids, colchicine, methotrexate, azathioprine, cyclosporine, chlorambucil, budesonide, pentoxifylline, nicotine, silymarin, vitamin E or pirfenidone in the preceding three months
* History of peripheral neuropathy
* Use of medications with significant drug-drug interactions with thalidomide
* History of Human Immunodeficiency Virus (HIV) positive status or Acquired Immunodeficiency Syndrome (AIDS)
* History of coexistent advanced malignancy
* History of coexistent severe cardiovascular disease
* History of coexistent severe renal disease
* History of current excessive or recent (within 6 months) alcohol use
* Any condition that, in the opinion of the investigators, would interfere with the patient's ability to complete the study safely or successfully
* History of thrombolytic events. Combination use with corticosteroids increases risk of deep vein thrombosis.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Lindor, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 4/6/2006 and 5/7/2009 at Mayo Clinic outpatient area.
Groups:
- Thalidomide: Patients with primary sclerosing cholangitis (PSC) who met with enrollment criteria were treated with 400 mg in the evening for a duration of 6 months
Period: Overall Study
Arm/Group | Thalidomide
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thalidomide
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase
Description: The primary outcome was the change in serum liver biochemical parameter levels after 6 months of thalidomide when compared to baseline values. This was to be analyzed using the nonparametric Wilcoxon signed rank test of significance. This was based on the non-normal distribution of serum hepatic biochemical parameters among patients with PSC and the continuous nature of these variables.
Time Frame: 6 months, baseline
Population: Analysis was not performed because participant did not complete the study due to adverse events.
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Thalidomide: Only one subject was enrolled, so study was terminated early.
Arm/Group | Thalidomide
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Toxicity and Tolerability
Description: Overall toxicity and tolerability were to be measured by the number of patients with development of neuropathy, increased liver biochemistries, drowsiness, dizziness and orthostatic hypotension.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Thalidomide
Number analyzed (Participants) | 0

3. Secondary Outcome: Mayo Risk Score
Description: The Mayo Risk Score estimates the survival probability of a patient with primary sclerosing cholangitis based on the following variables: age, bilirubin, albumin, AST and history of variceal bleeding.
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | Thalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Soluble Tumor Necrosis Factor - Alpha
Description: Assessment of effect from thalidomide on soluble tumor necrosis factor - alpha compared to baseline values were to be performed at study conclusion.
Time Frame: 6 months, baseline
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Thalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Thalidomide
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide (N=1)
hand pain (Nervous system disorders) | 1 (1)
loose stools (Gastrointestinal disorders) | 1 (1)
decreased appetite (Gastrointestinal disorders) | 1 (1)
aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
weight loss (General disorders) | 1 (1)
low blood pressure (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only one subject was enrolled, so study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No